CLINICAL TRIAL: NCT03436355
Title: Active School. A School-based Intervention to Increase Childrens Daily Physical Activity and Its Effect on Childrens Self-regulation
Brief Title: Active School. A School-based Intervention to Increase Childrens Daily Physical Activity Level.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Stavanger (Other)
Collaborators: Municipality of Stavanger (Unknown); Rogaland County Council (Unknown); Regional Research Fund, Norway (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Prosjektnr NSD: 38509
Record Dates: First submitted 2018-02-01; First posted 2018-02-19 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Physical Activity; Aerobic Fitness; Executive Function
Keywords: Behavioral; Physical activity; Intervention; School children
MeSH Terms: conditions — Motor Activity; Behavior | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical activity (Experimental): 60 minutes of daily physical activity (see intervention)
  Interventions: Behavioral: Physical activity

INTERVENTIONS:
Behavioral: Physical activity — The "Active school" study was a 10-month randomized controlled trial.The weekly interventions were 2×45 minutes physically active academic lessons, 5×10 minutes physically active breaks, and 5×10 minutes physically active homework.

SUMMARY:
This study seeks to explore whether increased physical activity in school affects children's executive function, aerobic Fitness and childrens self-regulation. The "Active school" study was a 10-month randomized controlled trial. The sample included 449 children (10-11 years old) in five intervention and four control schools. The weekly interventions were 2×45 minutes physically active academic lessons, 5×10 minutes physically active breaks, and 5×10 minutes physically active homework. Aerobic fitness was measured using a 10-minute interval running test. Executive function was tested using four cognitive tests (Stroop, verbal fluency, digit span, and Trail Making). A composite score for executive function was computed and used in analyses.

Self-regulation was measured by the Child Behavior Rating Scale.

ELIGIBILITY:
Inclusion Criteria:

* all children attending 5th grade at the included schools in Stavanger, Norway during the school-year 2014/2015.

Exclusion Criteria:

* not able to participate in daily physical activity and physical education and complete the cognitive tests.

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 449 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Inhibition | 8 months intervention
  Response inhibition was measured by Stroop Golden color-word test. Participants were naming the printed color of color words while suppressing the reading of the words. The measure was the number of words read in 45 Seconds.
Working memory | 8 months intervention
  Working memory was tested by the Wechsler Adult Intelligence Scale (WAIS)-IV-test, a forward and backward digit span, a test that measures working memory function. The measure was the length of the correct series of numbers repeated by the participant.
  was included
Cognitive flexibility | 8 months intervention
  Cognitive flexibility was tested by two tests. First the participants were asked to list all the animals they could think of in 60 seconds as fast as they could.The number of animals was the score. Second, participants performed the Trail Making test. This involves drawing a line connecting consecutive numbers from 1 to 25 as fast as possible. Then participants were drawing a similar line, connecting alternating numbers and letters in sequence, example: 1-A-2-B. Time to complete each "trail" was recorded.
Aerobic fitness | 8 months intervention
  Aerobic fitness was assessed by a 10-minute interval running test. The children ran back and forth between two lines placed 20 m apart, touching the ground behind the line with their hand every time they reversed direction.
  After 15 seconds, a teacher signaled stop and the children rested for 15 seconds before they once more ran for 15 seconds. This procedure lasted 10 minutes, and the running distance was the outcome measure.
Physical activity | 8 months intervention
  Physical activity was measured using accelerometry (ActiGraph GT1M/GT3X/GT3X+, LLC, Pensacola, Florida, USA).
  The children were asked to wear the accelerometer on the right hip for seven consecutive days, removing it only during water-based activities (e.g., swimming) and while sleeping. Data were considered valid if a child had at least two days with a wear time of ≥480 min/day accumulated between 06:00 and 24:00.

SECONDARY OUTCOMES:
Self-regulation | 8 months intervention
  Self-regulation was measured by the Child Behavior Rating Scale (CBRS). This is a teacher rating based on the Bronson Social Task and Skill Profile, designed to assess children's classroom goal-oriented behaviors and strategies used to regulate behavior in academic and social situations. The teacher report consisted of 10 items used to assess children's self-regulation in the classroom.

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Munthe, PhD, Study Chair — University of Stavanger

IPD SHARING:
Plan to Share IPD: Undecided
A plan to share data will be decided when all of the planned papers is published.

REFERENCES:
- [Result] Dyrstad SM, Kvalo SE, Alstveit M, Skage I. Physically active academic lessons: acceptance, barriers and facilitators for implementation. BMC Public Health. 2018 Mar 6;18(1):322. doi: 10.1186/s12889-018-5205-3. PMID 29510699
- [Result] Kvalo SE, Bru E, Bronnick K, Dyrstad SM. Does increased physical activity in school affect children's executive function and aerobic fitness? Scand J Med Sci Sports. 2017 Dec;27(12):1833-1841. doi: 10.1111/sms.12856. Epub 2017 Mar 16. PMID 28207976
- [Derived] Seljebotn PH, Skage I, Riskedal A, Olsen M, Kvalo SE, Dyrstad SM. Physically active academic lessons and effect on physical activity and aerobic fitness. The Active School study: A cluster randomized controlled trial. Prev Med Rep. 2018 Dec 28;13:183-188. doi: 10.1016/j.pmedr.2018.12.009. eCollection 2019 Mar. PMID 30656132